CLINICAL TRIAL: NCT04117919
Title: Pilot Study of Chinese Medicine Medicated Bath as Complementary Medicine for Mild to Moderate Plaque -Type Psoriasis Patient.
Brief Title: Psoriasis、Indigo Naturalis、Chinese Medicine Medicated Bath
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH107-REC2-182
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chinese medicine medicated bath (Experimental): we used the leaf of paper mulberry as chinese medicine medicated bath. Two packs per day ,and the period of treatment will be two month.
  Interventions: Drug: paper mulberry leaf; Drug: Triamcinolone (Encort-A) 0.1%15g/Tube
- control group (Active Comparator): Topical steroids
  Interventions: Drug: Triamcinolone (Encort-A) 0.1%15g/Tube

INTERVENTIONS:
Drug: paper mulberry leaf — Topical steroids+paper mulberry leaf The botanical origin of paper mulberry leaf is Broussonetia papyrifera (L.) Vent.
  Other Names: Triamcinolone (Encort-A) 0.1%15g/Tube; Encort-A
  Arms: chinese medicine medicated bath
Drug: Triamcinolone (Encort-A) 0.1%15g/Tube — only Topical steroids
  Other Names: Encort-A

SUMMARY:
Psoriasis is a chronic inflammatory skin disease. Plague-type psoriasis is the most common form of the disease, occurring in more than 80% of the cases. This type of psoriasis is characterized by sharply dermatcated, erythematous, scaling plagues that typically affect the elbows, knees, scalp, and trunk. Estimates of the prevalence of psoriasis was vary from 0.5% to 4.6%, with rate varying between countries and races. The prevalence of psoriasis was about 2% in Taiwan. The etiology of psoriasis remains unknown; however, current research mostly indicated that psoriasis was caused by multiple factors, and it was highly related to Th-17 immunal pathway.Treatment of psoriasis included topical therapy, phototherapy and systemic therapy. Although beneficial, those therapies often caused undesirable adverse effects. Traditional Chinese medicine is one of the most fuguently chosen alternative therapies in China and Taiwan, and psoriasis has been treated for centuries with topical and oral herbal prepations. Chinese medicine medicated bath is a characteristic therapy of Traditional Chinese medicine. It combines both hot bath and herbs to enhance absorption of the effective ingredients of herb. There were reports about the application of Chinese medicine medicated bath to treat psoriasis patients in China. We also used Chinese medicine medicated bath (Jing-Fu-Yau-Yu-Bau) as a complementary therapy of psoriasis patients for a long time in China Medical University Hospital. The patient felt well after using Jing-Fu-Yau-Yu-Bau. The component of Jing-Fu-Yau-Yu-Bau is paper mulberry leaf. The botanical origin of paper mulberry leaf is Broussonetia papyrifera (L.) Vent. It can clear heat, cool blood and relieve itching. Based on the 83 journal paper we searched on PubMed, there had been extracted a great deal of phenolics, terpenes and flavonoids from paper mulberry leaf that had antibacterial, antifungal, antioxidant and antineoplastic effects.

This is a single site, randomized, single-blind, controlled pilot study of Jing- Fu-Yau-Yu-Bau as a complementary therapy to treat mild to moderate plaque- type psoriasis during an 8-week period. We estimate to enroll 30 subjects (treatment group(N=15); controlled group(N=15)). We plan to investigate the efficacy and safety of Jing-Fu-Yau-Yu-Bau in Chinese subjects with mild to moderate plaque-type psoriasis.

DETAILED DESCRIPTION:
This is a single site, randomized, single-blind, controlled pilot study of Jing- Fu-Yau-Yu-Bau as a complementary therapy to treat mild to moderate plaque- type psoriasis during an 8-week period. We estimate to enroll 30 subjects (treatment group(N=15); controlled group(N=15)).

ELIGIBILITY:
Inclusion Criteria:

* 20-65 years,
* had a diagnosis of plaque-type psoriasis for ≥6 months,
* a Physician's Global Assessment (PGA) score of 2-3, <20% total body surface area (BSA) involvement, and a target plaque of ≥4 cm2.

Exclusion Criteria:

* non-plaque psoriasis,
* rebound/flare of chronic psoriasis,
* history of psoriatic arthritis,
* current drug-induced psoriasis,
* pregnant/nursing/planning pregnancy (men and women),
* used biologics within 3 months or 5 times the half-life,
* received phototherapy/systemic treatment within 4 weeks,
* topicals within 2 weeks,
* any systemic immunosuppressants within 4 weeks, -lithium/antimalarial/intramuscular gold within 4 weeks,
* tested positive for HIV/hepatitis B/C,
* had a history of alcohol/drug abuse,
* clinically-significant laboratory abnormality,
* sensitivity to Chinese herbs ,or allergy to leaf of paper mulberry.
* had skin wound or skin infection
* had current signs/symptoms of severe, progressive, or uncontrolled medical conditions, or were participating concurrently in an investigational study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-05 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-03 (Estimated)

PRIMARY OUTCOMES:
participants achieving either a major clinical response or partial clinical response defind by Psoriasis Area Severity Index(PASI) over the 8 weeks treatment period. | baseline to 8 weeks
  Psoriasis Area Severity Index(PASI) is usually measure the clinical activity diseases of psoriasis.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Man Cheng, Study Chair — China Medical University Hospital
Locations (1):
- No. 91, Xueshi Rd., North Dist., Taichung City 404, Taiwan (R.O.C.), Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No